CLINICAL TRIAL: NCT06667167
Title: A Prospective, Open-label, Single-arm, Phase II Study to Evaluate First Line Therapy for Extensive-stage Small Cell Lung Cancer (SCLC) Patients, Treated by Induction Carboplatin/etoposide/pembrolizumab Followed by Maintenance of Pembrolizumab/ Sacituzumab Govitecan
Brief Title: First Line Therapy for Extensive SCLC Patients, Treated with Chemo+Keytruda Followed by Keytuda+Trodelvy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nir Peled (Other)
Responsible Party: Sponsor-Investigator, Nir Peled, Head of Oncology, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240215 MISP_3475-F93
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: NSCLC (non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Etoposide; pembrolizumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Single Arm
  Interventions: Drug: Induction Carboplatin

INTERVENTIONS:
Drug: Induction Carboplatin — Induction phase of carboplatin+etoposide+pembrolizumab followed by maintenance of Pembrolizumab+sacituzumab govitecan
  Other Names: Carboplatin; Etoposide; Pembrolizumab; Sacituzumab Govitecan

SUMMARY:
Induction phase of carboplatin+etoposide+pembrolizumab followed by maintenance of Pembrolizumab+sacituzumab govitecan

DETAILED DESCRIPTION:
Patients with extensive small cell lung cancer, who are previously untreated for extensive disease, will receive induction chemotherapy of carboplatin and etoposide along with pembrolizumab. The patient will then receive maintenance therapy with pembrolizumab and sacituzumab govitecan.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of ES SCLC will be enrolled in this study.
2. The participant has not been previously treated with systemic therapy for ES SCLC (i.e., the disease is treatment naïve).

   Note: Participants previously treated for limited SCLC will be allowed with disease-free survival (DFS) of 6 months after completion of all treatment.
3. Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Note: Participants with asymptomatic brain metastases will be eligible. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Evaluation of ECOG is to be performed within 3 days prior to the first dose of study intervention.
8. Life expectancy >3 months.
9. Has adequate organ function as defined in the following table (Table 2). Specimens must be collected within 10 days prior to the start of study intervention.
10. A female participant is eligible to participate if she is not pregnant (refer to the Clinical Trials Facilitation and Coordination Group [CTFG] "Recommendations related to contraception and pregnancy testing in clinical trials", Appendix 5), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined by CTFG Recommendations (Appendix 5) or
    2. A WOCBP who agrees to follow the contraceptive guidance per CTFG Recommendations (Appendix 5) during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatments) after the last dose of study treatment.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Has received prior systemic anti-cancer therapy including biologic agents or investigational agents or an investigational device within 4 weeks prior to treatment initiation.
3. Has received prior radiotherapy, chemotherapy, or targeted small molecule therapy within 2 weeks of start of study intervention and have not recovered from AEs at the time of study entry (i.e., ≥Grade 2 is considered not recovered), or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system (CNS) disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
4. Have not recovered (i.e., ≥Grade 2 is considered not recovered) from AEs due to a previously administered agent.

   Note: participants with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study.
5. Have previously received topoisomerase 1 inhibitors.
6. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed. (Refer to Section 5.5 for information on COVID-19 vaccines).
7. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.
8. Has a known hypersensitivity to any of the study treatments, their metabolites, or formulation excipients.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
11. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid).
13. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
14. Has an active infection requiring systemic therapy.
15. Has an active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months of enrollment.
16. Have a history of, or active hepatitis B virus (HBV) or hepatitis C virus (HCV).

    Note: Testing for Hepatitis B or C is not required unless mandated by local health authority.
17. Has not adequately recovered from major surgery or has ongoing surgical complications.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.
22. History of HIV infection. Note: HIV testing is not required unless mandated by local health authority.

    -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Hypothesis: The addition of SG to pembrolizumab in the post induction phase of the KEYNOTE-604 regimen will improve PFS of participants with first-line ES SCLC.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study the data will be published including relevant IPD